CLINICAL TRIAL: NCT04462666
Title: Oral Huzhang Granules for Acute Gouty Arthritis: Protocol for a Randomized, Double-blind, Multicenter Clinical Trial
Brief Title: Oral Huzhang Granules for Acute Gouty Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020024
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Gouty Arthritis
Keywords: Gouty arthritis; Randomized controlled trial; Huzhang granule; Traditional Chinese medicine
MeSH Terms: conditions — Arthritis, Gouty | interventions — Etoricoxib; Drug Contamination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HZG intervention (Experimental): During the 5-day treatment period, participants in the Experimental group will receive 10 sacks of experimental granules. They will be instructed to take two sacks per day, one in the morning and one in the evening, in approximately 30 minutes after the meal.. The placebo etoricoxib will also be taken daily in the morning for 5 days.
  Interventions: Drug: Huzhang granule; Drug: Etoricoxib Placebo
- Etoricoxib intervention (Active Comparator): During the 5-day treatment period, participants in the Etoricoxib group will receive 5 Etoricoxib capsules. They will be instructed to take one capsule per day in the morning, at approximately 30 minutes after the meal. The placebo HZKL will also be taken daily in the morning for 5 days.
  Interventions: Drug: Etoricoxib; Drug: Huzhang granule Placebo
- Placebo intervention (Placebo Comparator): During the 5-day treatment period, participants in the Placebo group will receive 10 sacks of placebo HZG. They will be instructed to take two sacks per day, one sack in the morning and one in the evening, at approximately 30 minutes after the meal. And the placebo etoricoxib also be taken daily in the morning for 5 days.
  Interventions: Drug: Huzhang granule Placebo; Drug: Etoricoxib Placebo

INTERVENTIONS:
Drug: Huzhang granule — Empty the content of one sachet into a mug, add 50ml warm water, stir until dissolved, add another 50ml hot water. Consume and complete all 100ml liquid mixture as a single dosage.
  Other Names: Chinese Herbal Medicine
  Arms: HZG intervention
Drug: Etoricoxib — take one capsule per day in the morning, at approximately 30 minutes after the meal.
  Other Names: Chemical drug
  Arms: Etoricoxib intervention
Drug: Huzhang granule Placebo — Empty the content of one sachet into a mug, add 50ml warm water, stir until dissolved, add another 50ml hot water. Consume and complete all 100ml liquid mixture as a single dosage.
  Other Names: Chinese Herbal Medicine
  Arms: Etoricoxib intervention; Placebo intervention
Drug: Etoricoxib Placebo — take one capsule per day in the morning, at approximately 30 minutes after the meal.
  Other Names: Chemical drug
  Arms: HZG intervention; Placebo intervention

SUMMARY:
We designed this study as a double-blind, randomized, controlled clinical trial. The aim of the study is to evaluate the clinical efficacy, safety and control of recurrence rate of acute gouty arthritis

DETAILED DESCRIPTION:
Gout is a recurrent chronic inflammatory disease caused by monosodium urate (MSU) crystal . Acute gouty arthritis (GA) is the most common first symptom of gout. With the progress of the disease, the frequency of acute attack increases, and joint destruction may occur. The prevalence of hyperuricemia in China was about 13.3%, and the pooled prevalence of gout was 1.1%. Repeated attacks of GA seriously affect the quality of life, resulting in huge economic costs and mental stress. Due to inadequate prevention and treatment, the target of healing gout is often not achieved. In GA, TCM has shown satisfactory therapeutic effect with less adverse effects and minimal toxicity. Huzhang granule (HZG), a Chinese herbal prescription, is a compound preparation with twelve ingredients which has been used in the clinical treatment of gout for over 30 years at the Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of TCM.Therefore，this double-blind, randomized, controlled clinical trial. will provide high-quality clinical evidences for evaluating the clinical efficacy, safety and control of recurrence rate of Huzhang granule ，a representative prescription for the treatment of acute gouty arthritis , in the treatment of GA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute gout arthritis as defined by the American College of Rheumatology 1977 preliminary criteria;
* Male or non-pregnant, non-nursing female;
* 18-70 years of age;
* Gout attack less ≤48 hours;
* In the week before this observation, non-steroidal anti-inflammatory drugs and analgesic drugs and drugs affecting uric acid metabolism were not taken;
* Subjects capable of giving informed consent;

Exclusion Criteria:

* failing to meet the diagnostic criteria;
* Evidence of uncontrolled concomitant cardiovascular, nervous system,hepatic or gastrointestinal disease. Potential participants who have active concomitant disease can only be eligible after discussion and agreement with the treating medical team;
* the patient is in critical condition and it is difficult to evaluate the effectiveness and safety of the clinical observation;
* severe deformity, stiffness and labor loss of patients with advanced arthritis;
* known allergic to the drug used in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | Up to 5 days after treatment
  Visual Analogue Score is an often-used tool to measure subjective phenomena, which has shown good reliability and validity in terms of assessment of pain. In the clinical study of acute gout attack，it can be used as a tool to measure the degree of pain from 0 to 100 mm (with 0 being no pain and 100 being maximum pain)

SECONDARY OUTCOMES:
Likert scales for the assessment of joint tenderness and swelling | Up to 5 days after treatment
  Likert scales for the assessment of joint tenderness and swelling is evaluate the inflammatory response and the degree of injury of the joint.Scores range from 1-5, a higher score indicating a severe symptoms on a participant's joint
symptom relief time | Up to 5 days after treatment
  Symptom relief time is the time when joint pain feels relieved
36-Item Short Form Survey | Up to 5 days after treatment
  36-Item Short Form Survey is a health status profile originally designed to measure eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  Scoring the 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key in a given table. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. another lists the items averaged together to create each scale. Items that are left blank (missing data) are not taken into account when calculating

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Shanghai Yueyang Integrated Medicine Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou M, Hua L, Wang YF, Chen ST, Yang CM, Zhang M, Li X, Li B. Oral Huzhang granules for the treatment of acute gouty arthritis: protocol for a double-blind, randomized, controlled trial. Trials. 2022 Apr 1;23(1):248. doi: 10.1186/s13063-022-06188-x. PMID 35365187